CLINICAL TRIAL: NCT04582370
Title: Impact of Theater Experience on Older Adults Living in Retirement Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, Director of Research, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000526106
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Aging
Keywords: Older adults; Theater; Physical functioning; Emotional stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theater program (Experimental): The design of the 10-week theater program is based on the principles of acting as written and practiced by Constantin Stanislavski in his revolutionary text on acting: "An Actor Prepares" [Stanislavsky C, 1989]. The exercises target concentration, voice, physical skills, emotion memory, observation, and dramatic analysis and include 3 components: 1. Preparation for the Actor (which involves relaxation , collaboration, movement, posture, and vocality; 2. Learning the Components of the Repeatable Acting Process (which involves physicality, attention, and concentration); and 3. Synthesizing Components into Characterization (which involves creativity and emotional expression).
  Each of these components will be addressed during each of 20 sessions through the use of group warm ups, group ensemble exercises, and group recitations. Participants will perform physical, mental, and emotional exercises similar to those given to beginning acting students in traditional theater schools.
  Interventions: Behavioral: theater program
- Wait-list control (No Intervention): During the study period, the control group will not receive any type of intervention. However, they will be offered the same theater program experience after the primary data collection period ends.

INTERVENTIONS:
Behavioral: theater program — 10-week theory-based theater program designed to improve their physical functioning and reduce emotional stress.
  Arms: Theater program

SUMMARY:
Theater is a complex, multi-component performing art. On stage, actors not only need to memorize the script, but also be able to portray emotion and feeling through movement and move in whichever manner is deemed appropriate by the script. Acting therefore requires as much movement as it does vocalization. As training exercises in theater naturally involve boosting physical, cognitive and affective function, and social relationships, theater experience can be used to promote health and wellness. Over the last two decades, there has been an increase in the use of theater to promote health and wellness among older adults.

Thus, the overall aim of this project is to evaluate the therapeutic benefits of a 10-week theory-based theater program on physical functioning and emotional stress among older adults.

Hypothesis #1: Older adults residing in subsidized housing who participate in a theory-based theater program will demonstrate better physical functioning, and reduction in emotional stress than wait-list controls at the conclusion of a 10-week theater program.

Hypothesis #2: The positive impact of the theater program on the residents' improved physical functioning and stress level will be maintained at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 62 or older living in HUD-subsidized housing
2. Residence in a subsidized apartment for at least one year.
3. Able to carry on a daily conversation with or without hearing aids
4. Intact cognition as indicated by a score of greater than 5 on the Short Portable Mental Status Questionnaire (SPMSQ)
5. Ambulatory with or without aids, as the outcome measures require participants to perform static and dynamic balance, and walking activities.

Exclusion Criteria:

1. Visual impairment that cannot be corrected with assistive devices
2. Diagnosis of progressive neurodegenerative disorders (self-report)

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Timed Up-and-Go | baseline
  The "timed Up-and-Go" (TUG) is a composite measure of functional mobility, including lower extremity power, balance, gait, and fall risk. Measured in absolute time (seconds), where lower time is a better score.
Timed Up-and-Go | immediately post-intervention
  The "timed Up-and-Go" (TUG) is a composite measure of functional mobility, including lower extremity power, balance, gait, and fall risk. Measured in absolute time (seconds), where lower time is a better score.
Timed Up-and-Go | 3-month follow up
  The "timed Up-and-Go" (TUG) is a composite measure of functional mobility, including lower extremity power, balance, gait, and fall risk. Measured in absolute time (seconds), where lower time is a better score.

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form | baseline
  The Medical Outcomes Study Short Form, version 2 (SF-36v2) is a 36 item patient reported outcome measure of health-related quality of life in 8 different domains. Scores range from 0 to 100, with high scores indicating more positive health.
Medical Outcomes Study Short Form | immediately post-intervention
  The Medical Outcomes Study Short Form, version 2 (SF-36v2) is a 36 item patient reported outcome measure of health-related quality of life in 8 different domains. Scores range from 0 to 100, with high scores indicating more positive health.
Medical Outcomes Study Short Form | 3-month follow up
  The Medical Outcomes Study Short Form, version 2 (SF-36v2) is a 36 item patient reported outcome measure of health-related quality of life in 8 different domains. Scores range from 0 to 100, with high scores indicating more positive health.
2-minute step test | baseline
  The 2-minute step test (TMST) is a field test of exercise tolerance where the participant steps in place for 2 min. The higher the number repetition indicates better performance.
2-minute step test | immediately post-intervention
  The 2-minute step test (TMST) is a field test of exercise tolerance where the participant steps in place for 2 min. The higher the number repetition indicates better performance.
2-minute step test | 3-month follow up
  The 2-minute step test (TMST) is a field test of exercise tolerance where the participant steps in place for 2 min. The higher the number repetition indicates better performance.
30-sec chair stand test | baseline
  The 30-sec chair stand test (30CST) is a measure of lower extremity power and functional mobility. The participant stands up from a chair and sits back down as many times as possible in 30 sec. The higher the number repetition indicates better performance.
30-sec chair stand test | immediately post-intervention
  The 30-sec chair stand test (30CST) is a measure of lower extremity power and functional mobility. The participant stands up from a chair and sits back down as many times as possible in 30 sec. The higher the number repetition indicates better performance.
30-sec chair stand test | 3-month follow up
  The 30-sec chair stand test (30CST) is a measure of lower extremity power and functional mobility. The participant stands up from a chair and sits back down as many times as possible in 30 sec. The higher the number repetition indicates better performance.
Berg Balance Scale | baseline
  The Berg Balance Scale (BBS) is a 14-iten test that measures function mobility and balance. Scores range from 0 to 56, with higher scores indicating better balance.
Berg Balance Scale | immediately post-intervention
  The Berg Balance Scale (BBS) is a 14-iten test that measures function mobility and balance. Scores range from 0 to 56, with higher scores indicating better balance.
Berg Balance Scale | 3-month follow up
  The Berg Balance Scale (BBS) is a 14-iten test that measures function mobility and balance. Scores range from 0 to 56, with higher scores indicating better balance.
Grip strength | baseline
  Hand-grip strength is a quantitative measure of upper extremity strength. Higher values indicated more strength.
Grip strength | immediately post-intervention
  Hand-grip strength is a quantitative measure of upper extremity strength. Higher values indicated more strength.
Grip strength | 3-month follow up
  Hand-grip strength is a quantitative measure of upper extremity strength. Higher values indicated more strength.
Emotional stress | baseline
  Emotional stress will be assessed via cortisol levels obtained from hair samples analyzed via immunoassay. Typical values range from 2 to 200 pg/mg, with higher levels indicating higher chronic stress.
Emotional stress | immediately post-intervention
  Emotional stress will be assessed via cortisol levels obtained from hair samples analyzed via immunoassay. Typical values range from 2 to 200 pg/mg, with higher levels indicating higher chronic stress.
Emotional stress | 3-month follow up
  Emotional stress will be assessed via cortisol levels obtained from hair samples analyzed via immunoassay. Typical values range from 2 to 200 pg/mg, with higher levels indicating higher chronic stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stanislavsky C. An Actor Prepares. New York: Routledge; 1989.
- [Derived] Kirklin K, Qu H, Mayor E, Lowman JD, Gao J, Edwards L, Li P, Yuen HK. The "Method of Physical Action" in Theatre Training Improves Balance and Reduces Fall Risk in Older Adults Living in Subsidized Housing: A Randomized Controlled Trial. Innov Aging. 2025 May 6;9(6):igaf046. doi: 10.1093/geroni/igaf046. eCollection 2025. PMID 40600024